CLINICAL TRIAL: NCT06871683
Title: ClotTriever® Thrombectomy System Use-Result Survey in Japan
Status: Enrolling by invitation | Type: Observational
Sponsor: Inari Medical (Industry)
Collaborators: Vorpal Technologies (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24-001
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full Analysis Population: All subjects who the survey device entered their vasculature.
  Interventions: Device: ClotTriever® Thrombectomy System

INTERVENTIONS:
Device: ClotTriever® Thrombectomy System — ClotTriever® Thrombectomy System use for treatment of patients with deep vein thrombosis with acute severe symptoms.

SUMMARY:
The objective of this survey is to determine the safety and efficacy of the ClotTriever Thrombectomy System under daily clinical practice after marketing approval in Japan.

This device was designated as a subject of use results evaluation at the time of application for manufacturing and marketing approval.

ELIGIBILITY:
This is an all-comers survey of all patients treated with ClotTriever® Thrombectomy System in Japan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with deep vein thrombosis with acute severe symptoms (excluding postthrombotic syndrome) for whom the ClotTriever® Thrombectomy System was used. Patients will be enrolled until at least 100 subjects complete the follow-up period through 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events | Through 30 days post index procedure.
  Rate of Major Adverse Events [All-cause mortality, Major bleeding, New symptomatic Pulmonary Embolism (PE) documented by Computed Tomography Pulmonary Angiography (CTPA), Rethrombosis of a Target Venous Segment].
Technical Success | During the index procedure
  Thrombus residual volume assessed by the the treating physician using pre- and post-procedure venography to evaluate the success of thrombus removal.

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Chiba University Hospital, Chuo, Chiba
  - Ota Memorial Hospital, Ōta, Gunma
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Asahikawa Medical Hospital, Asahikawa
  - Asahi General Hospital, Chiba
  - Nozaki Tokushukai Hospital, Daitō
  - Shonan Kamakura, Kanagawa
  - Kyoto Katsura Hospital, Kyoto
  - Nara City Hospital, Nara
  - Mie University, Tsu